CLINICAL TRIAL: NCT02268578
Title: Efficacy of Transcranial Direct Current Stimulation for Treating Working Memory Dysfunction and Depression For Patients With Temporal Lobe Epilepsy
Brief Title: Efficacy of TDCS for Treating Working Memory Dysfunction and Depression in Temporal Lobe Epilepsy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Epilepsy Foundation (Other); American Epilepsy Society (Other); American Academy of Neurology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S12-03395
Record Dates: First submitted 2014-10-02; First posted 2014-10-20 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Epilepsy
Keywords: Transcranial Direct Current Stimulation; TDCS; Memory Dysfunction; Depression
MeSH Terms: conditions — Epilepsy; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial Direct Current Stimulation (Active Comparator): Subjects will receive a total of 5 sessions on consecutive days. During each session, 2 mA of tDCS will be applied for 20 minutes over the left DLPFC (active or sham). The electrodes will have the size of 35cm2 each. Direct current will be transferred by a saline-soaked pair of surface sponge electrodes and delivered b y a specially developed, battery driven, constant current stimulator with a maximum output of 2mA.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham TDCS (Sham Comparator): For sham-controlled tDCS subjects, the same montage will be used; however current will be applied for only 30 seconds - this is a reliable method of sham stimulation as sensations arising from tDCS treatment occur only at the beginning of application as also demonstrated by a randomized study (Gandiga et al. 2006).
  Interventions: Procedure: Sham Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — 2mA tDCS
  Arms: Transcranial Direct Current Stimulation
Procedure: Sham Transcranial Direct Current Stimulation — Transcranial Direct Current Stimulation is administered but at 0mA
  Arms: Sham TDCS

SUMMARY:
Memory difficulty ranks among the most common complaints for patients with temporal lobe epilepsy. While these cognitive problems may affect quality of life more than seizure frequency, no effective therapy exists. Transcranial Direct Current Stimulation (tDCS) is a method of safe, noninvasive, and painless brain stimulation delivering low intensity direct current through scalp electrodes to modulate brain activity. Several recently published studies demonstrate the enhancement of working memory and mood with stimulation of the frontal region of the brain. Furthermore, tDCS has never been reported to have induced a seizure. The aim of our study is to determine whether real tDCS can improve memory function and mood. The investigators are enrolling patients with well-controlled temporal lobe epilepsy who have not undergone brain surgery.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a powerful technique to modulate brain activity:

TDCS is based on the application of a weak direct current to the scalp that flows between two relatively large electrodes-anode and cathode. During tDCS, low amplitude (1-2 mA), constant currents are applied via the scalp electrodes and penetrate the skull to enter the brain. Although there is substantial shunting of current in the scalp, sufficient current penetrates the brain to modify the trans-membrane neuronal potential as shown by two recent modeling studies (Miranda et al. 2006; Wagner et al. 2007a), and thus influence the level of excitability and modulate the firing rate of individual neurons. When tDCS is applied for a sufficient duration, cortical function can be altered beyond the stimulation period (Nitsche and Paulus 2001) and the direction of the cortical excitability changes depends on current orientation.

Several well-conducted animal studies on the effects of tDCS dating back to the 1950s and 60s showed that tDCS is a powerful technique to modulate brain function. These studies demonstrated that polarizing currents applied to the surface of the brain result in a modulation of the cortical activity. Surface anodal polarization of the cortex increases spontaneous unit discharges (Burns 1954; Creutzfeld et al. 1962) and initiates paroxysmal activity (Goldring and O'Leary 1951), whereas cathodal polarization generally depresses these events. Furthermore, low-level surface polarization facilitates acquisition of learned motor responses and induces prolonged changes in patterns of evoked cortical unit discharges (Bindman et al. 1964). Finally, Purpura et al. (1964), studying pyramidal tract cells from cats, showed that prolonged periods of polarization may produce progressive membrane and post-synaptic potential changes as well as after-effects (Purpura and McMurtry 1965).

Based on this evidence, recent human studies have been performed and collectively have shown that motor cortex (M1) stimulation with tDCS changes motor cortex excitability depending on the stimulation polarity: while anodal stimulation increases cortical excitability, cathodal stimulation decreases it (Nitsche et al. 2003; Nitsche and Paulus 2000; Nitsche and Paulus 2001). Similar modulatory effects have also been described in the visual cortex (Antal et al. 2004; Antal et al. 2001). A recent tDCS study has shown that anodal tDCS of the primary motor cortex not only affects cortical activity, but induces significant changes on thalamic activity (Lang et al. 2005). It should be noted that application of tDCS in humans has advanced significantly in the last 10 years and it is therefore different from the human application used in the '60s and '70s (Wagner et al. 2007b)

Furthermore, tDCS offers several advantages as compared with other techniques of noninvasive brain stimulation (i.e., repetitive transcranial magnetic stimulation (rTMS)): (1) small size of the electrodes and stimulator, thus allowing portable use for instance to be used at home, (2) simple and non-expensive technique that can easily be translated for use in clinical practice, (3) long-lasting effects - the modulatory effects of tDCS last longer as compared to rTMS - for instance, 13 minutes of stimulation changes brain excitability for up to 2 hours (Nitsche and Paulus 2001), and (4) more easily blinded with sham tDCS in the setting of clinical trials (Gandiga et al 2006)

Prefrontal stimulation has been shown to enhance cognitive function:

There have been several recently published studies demonstrating the enhancement of working memory when tDCS stimulation is applied to the dorsal lateral prefrontal cortex. Fregni et al (2005) studied 15 normal subjects. The patients performed a three -back working memory task during active anodal (stimulatory) tDCS of the left dorsolateral prefrontal cortex (left DLPFC), sham stimulation over the left DLPFC, cathodal (inhibitory) stimulation of the left DLPFC, or anodal stimulation over the primary motor cortex (M1). The results of this study showed a significant improvement in working memory as indexed by task accuracy after active anodal tDCS of the left DLPFC. The other conditions of stimulation-including sham tDCS, anodal tDCS of left DLPFC, or anodal tDCS of M1-did not result in a significant task performance change. Similarly, Boggio et al (2007) have also found significant improvement in affective go-no-go task performance in patients with severe depression after treatment with anodal tDCS to the left DLPFC independent of the degree of mood enhancement after 10 consecutive days of tDCS.

Conversely, there has been some evidence that cathodal inhibition of the right DLPFC enhances working memory performance in the same task in depressed patients (Bermpohl et al 2006). Together these studies suggest that the increased activity of the left DLPFC-whether directly through anodal stimulation or indirectly through cathodal inhibition of the right DLPFC-is responsible for improvement in working memory performance.

Transcranial direct current stimulation (tDCS) has a significant antidepressant effect: Modulation of prefrontal cortex with anodal tDCS is associated with a significant improvement in depression. Initially a preliminary, randomized, controlled and double blind trial in which the effects of five days of anodal stimulation of the left DLPFC in 10 patients with major depression was investigated. All patients tolerated tDCS without complications. At the end of treatment, there were 4 treatment responders in the active group versus no responders in the sham group. The patients who received active stimulation had a significant decrease in the Hamilton Depression Rating Scale (HDRS) and Beck Depression Inventory (BDI) scores compared to baseline which was not observed in patients that received sham stimulation (Fregni et al. 2006b).

In a follow-up, parallel-group, double-blind clinical trial with 40 patients with major depression, patients were washed-out of their medications and randomized into three groups of treatment: anodal tDCS of the left DLPFC (active group); anodal tDCS of the occipital cortex (active control group) and sham tDCS (placebo control group). tDCS was applied for 10 sessions during a 2-week period. Mood was evaluated by a blinded rater using the HDRS and BDI. The treatment was well tolerated with minimal side effects that were distributed equally across all treatment groups. This study showed significantly larger reductions in depression scores after left DLPFC tDCS (HDRS reduction of 40.4% (±25.8%)) as compared to occipital (HDRS reduction of 21.3% (±12.9%)) and sham tDCS (HDRS reduction of 10.4% (±36.6%)). The beneficial effects of tDCS in the DLPFC group persisted for 1 month after the end of treatment (Boggio et al. 2008).

Similarly, in another longitudinal study on depression by Rigonatti et al (2008), serial applications of anodal (stimulatory) tDCS applied to the prefrontal cortex (10 sessions of 2 mA each) had a similar effect on reducing depressive symptoms as measured by Beck Depression Inventory scores as fluoxetine even 6 weeks after treatment. However, the effects of tDCS were more immediate than that of fluoxetine19.

In summary, tDCS of the left DLPFC seems to be able to induce significant positive affective and cognitive improvements in normal patients and patients with significant depression. We will therefore in this proposal test whether prolonged prefrontal stimulation is associated with clinically meaningful changes in affective and cognitive function without worsening epileptiform activity or seizure frequency. The results of this pilot study will have a significant clinical impact for the treatment of the neuropsychiatric comorbidities of patients with temporal lobe epilepsy.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18-70 years
2. diagnosis of temporal lobe epilepsy, with seizure focus defined by seizure semiology, EEG, MRI Brain, PET and/or ictal and interictal SPECT.
3. Must have a stable seizure frequency in the two (2) months prior to enrollment, as verified by the patient's seizure log and/or clinic notes and without recent antiepileptic medication changes.
4. Must score above 22/30 on the Montreal Cognitive Assessment (MoCA).
5. Must be able to provide informed consent.

Exclusion Criteria:

1. Patient has a progressive or unstable neurological or systemic disease
2. Patient has an ictal focus over the F3 or F4 (DLPFC) field
3. Patient has a history of severe depression, as determined by a screen inventory test such as the Beck Depression Inventory or a psychiatrist
4. Patient has a history of severe traumatic brain injury or prior brain surgery with skull defect
5. Contraindictations to tDCS, including metal in the head or implanted brain medical devices
6. Pregnancy
7. Any implanted electrical medical device, including pacers and implanted cardiac defibrillators
8. History of schizophrenia, schizoaffective disorder, other psychosis, rapid-cycling bipolar illness, alcohol/drug abuse within the past year
9. History of dementia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in EEG Power | Visits 1, 5, 6 & 7 over 5 weeks

SECONDARY OUTCOMES:
Cognitive Tests | Visits 1, 5, 6 & 7 over 5 weeks
  RAVLT Digits forward and backward testing Letter and Number Sequencing Visuospatial working memory and executive function tests

CONTACTS AND LOCATIONS:
Overall Officials: Anli Liu, MD, Principal Investigator — NYU Langone Health
Locations (1):
- Neurology, New York, New York, United States